CLINICAL TRIAL: NCT04295668
Title: PAPRIKA - Patients Empowerment for Major Surgery Preparation @Home
Acronym: PAPRIKA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Anael Barberan-Garcia, Principal investigator, Hospital Clinic of Barcelona
Other Study IDs: HCB/2019/1030
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cancer; Surgical Procedure, Unspecified
Keywords: Prehabilitation; Exercise training; Physical activity; Nutrition; Cognitive behavioural therapy; Smoking cessation; eHealth
MeSH Terms: conditions — Neoplasms; Motor Activity; Smoking Cessation | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual care: A contemporaneous control group of patients was build using propensity score matching (PSM) methodologies taking into account the following matching variables: type of surgery, age, sex, American Society of Anesthesiologists Index (ASA) and adjusted morbidity groups (GMA) grading.
  Interventions: Behavioral: Usual care
- Prehabilitation: Prospective sample of risk patients who are candidates for major surgery attended in the outpatient offices of the Hospital Clínic de Barcelona.
  Inclusion criteria: i) American Society of Anesthesiologists Index (ASA) 3-4; and / or, ii) age ≥ 75 years; and / or iii) major aggressive surgery; and, iv) solid organ transplant candidate.
  Exclusion criteria: i) Non-elective surgery; ii) Known metastatic disease before surgery; iii) Unstable respiratory or heart disease; or, iv) Locomotive or cognitive limitations that prevent adherence to the program.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Usual care — The preoperative standard measures consist of physical activity recommendation and advice on both smoking cessation and alcohol intake reduction. Moreover, in patients presenting with anemia, the anesthesiologists will assess its etiology and treat it accordingly, and nutritional intervention will be performed by a registered dietitian in to those patients at risk of malnutrition (Malnutrition Universal Screening Tool ≥2).
  Groups: Usual care
Behavioral: Prehabilitation — i) Exercise training: Ambulatory exercise training sessions with two main components, namely: high-intensity endurance exercise training and strength muscular training.
  ii) Promotion of physical activity: Pedometer-based program using a physical activity tracker linked to a mobile app.
  iv) Nutritional optimization: Recommendations of a healthy balanced diet or adapted to their digestive symptoms. Daily amount of protein intake will be close to 2 g•Kg-1•day-1.
  iv) Smoking cessation: Use of both cognitive behavioral intervention and pharmacological therapy by varenicline or nicotine replacement therapies.
  v) Cognitive behavioral therapy: Weekly group sessions conducted by a clinical health psychologist, including psychoeducation, motivational and behavioral change, self-efficacy and adherence enhancement, coping strategies acquisition and patient empowerment.
  Groups: Prehabilitation

SUMMARY:
PAPRIKA establishes a technologically enabled and personalized prehabilitation and follow-up after surgical intervention program for patients undergoing elective major surgery Program creates close collaboration between the medical environment and the patients empowering them to co-create their own care.

It is at the first stage aimed to high-risk patients undergoing major surgery. Better condition before the surgery is proved to reduce the perioperative complications and to improve patients' health-related quality of life while cutting the associated costs. The concept integrates short-term (average 4 weeks) preoperative interventions including endurance training, promotion of physical activity and nutritional and psychological support. Interventions are planned both at community and at hospital reducing unnecessary interactions between patients and tertiary care.

PAPRIKA tackles three major drivers: i) human perspective ii) organizational challenges and iii) technical aspects. The project is based on previous experience on prehabilitation and the already refined service using design thinking methodologies. It will be also based on the proven reduction of associated costs for the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years old and/or American Society of Anesthesiologist (ASA) index 3-4 and/or highly aggressive surgery or solid organ transplantation.

Exclusion Criteria:

* Non-elective surgery; metastatic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective sample of risk patients who are candidates for major surgery attended in the outpatient offices of the Hospital Clínic de Barcelona.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Duration of the initial hospitalization for surgery
  Number of postoperative complications during the initial hospitalization for surgery
Hospital length of stay | Duration of the initial hospitalization for surgery
  Number of days of hospital length of stay during the initial hospitalization for surgery
Severity of postoperative complications | Duration of the initial hospitalization for surgery
  Severity of postoperative complications during the initial hospitalization for surgery using the Clavien-Dindo classification

SECONDARY OUTCOMES:
Hospital readmissions at 30 days | From initial hospital discharge to 30 days follow-up
  Number of postoperative complications during a 30-day period after surgery
Emergency room visits at 30 days | From initial hospital discharge to 30 days follow-up
  Number of emergency room visits during a 30-day period after surgery
Surgical reinterventions at 30 days | From initial hospital discharge to 30 days follow-up
  Number of surgical reinterventions during a 30-day period after surgery
Mortality at 30 days | From initial hospital discharge to 30 days follow-up
  Number of exitus during a 30-day period after surgery

OTHER OUTCOMES:
Six-minute walk test | At program inclusion and at program discharge (on average at 6 weeks)
  Distance covered during the six-minute walk test
Physical activity | At program inclusion and at program discharge (on average at 6 weeks)
  Physical activity measured by the Yale Physical Activity Survey (YPAS) (range 0 to 142; the lowest the worst)
Psycho-emotional status | At program inclusion and at program discharge (on average at 6 weeks)
  Psycho-emotional status measured by the Hospital Anxiety and Depression (HAD) scale (range 0-21; the highest the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Roca, Prof, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided